CLINICAL TRIAL: NCT03101345
Title: Assessment of Nutrition on Brain Energy Metabolism: Measurement of High Energy Phosphate Metabolites by 31-phosphorous Magnetic Resonance Spectroscopy.
Brief Title: High Energy Phosphate Metabolites in Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16.19.CLI
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nutrition product (Other): Peptamen® 1.5 Vanilla, orally administration
  Interventions: Other: Peptamen® 1.5 vanilla

INTERVENTIONS:
Other: Peptamen® 1.5 vanilla — Administration orally

SUMMARY:
The objective of this research project is to determine the impact on brain HEP metabolites and fluxes of an oral consumption of a commercially available nutrition product (Peptamen® 1.5 vanilla) in healthy volunteers.

Therefore, we intend to perform 31P-MRS before and after oral intake of the nutrition product.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18-45 years
* Healthy, based on the medical screening visit
* Normal BMI for age (18.5-25.0 kg/m2)
* Able to understand and to sign a written informed consent prior to trial entry
* Informed consent signed

Exclusion Criteria:

* Known type 1 or type 2 diabetes, on anamnesis
* Family history of type 2 diabetes (parents)
* Any other metabolic disease possibly impacting the postprandial glucose and insulin response (on anamnesis, to the opinion of the medical expert)
* Malabsorptive disorders including but not limited to pancreatitis, Crohn's disease, etc
* Any history of neurological / psychological disease (meningitis, epilepsy), to the opinion of the investigator
* Claustrophobia
* Hearing disorders
* Any medication impacting dietary fat absorption and metabolism like statins, bile acid sequestrants, lipid lowering medications, or fibrates , to the opinion of the medical expert
* Pregnancy (on anamnesis) and/or lactation
* Having any metallic, electronic, magnetic, or mechanical implants, devices, or objects, for safety reason linked to magnetic field exposure (MRS):

  * Aneurysm clip(s)
  * Cardiac pacemaker
  * Implanted cardioverter defibrillator (ICD)
  * Electronic implant or device
  * Magnetically-activated implant or device
  * Neurostimulation system
  * Spinal cord stimulator
  * Cochlear implant or implanted hearing aid
  * Insulin or infusion pump
  * Implanted drug infusion device
  * Any type of prosthesis or implant
  * Artificial or prosthetic limb
  * Any metallic fragment or foreign body
  * Hearing aid
  * Other implant
* Subject injured by a metallic object or foreign body
* History of cancer within the past year
* Allergy or intolerance to any food or compound used
* Currently following a strict exercise program (minimum three times per week) in order to either lose weight, gain muscle or reach competition standards for a chosen sport
* Currently participating or having participated in a clinical trial during the past month
* Subjects not willing and/or not able to comply with scheduled visits and the requirements of the research protocol. Subject having a hierarchical link with the investigator or co-investigators.
* Subject who cannot be expected to comply with the research protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
31P metabolites | 31P metabolites and fluxes will be measured during one hour 2 times, one before product intake (control) and the second one 45 min after product intake"
  The change in concentration of brain 31P metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Principal Investigator — Société des Produits Nestlé (SPN)
Locations (1):
- Metabolic Unit, Clinical Development Unit, Nestec, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No